CLINICAL TRIAL: NCT02090907
Title: Effects of Levothyroxine on Endothelial Function of Patients With Subclinical Hypothyroidism
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Nasmi Niknam, Dr., Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 392349
Record Dates: First submitted 2014-03-12; First posted 2014-03-18 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Subclinical Hypothyroidism
Keywords: Subclinical hypothyroidism; Atherosclerosis; Cardiovascular disease; Endothelial function; Prevention
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases | interventions — Thyroxine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levothyroxin (Experimental): In the treatment group, daily doses of 100 mg of Levothyroxine will be administered every morning, half an hour before breakfast.
  Interventions: Drug: Levothyroxine
- Placebo (Placebo Comparator): In the placebo group treatment regimen and advices are identical to that of the treatment group, except for using a pharmacologically neutral agent, with complete resemblance to the real treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levothyroxine
  Arms: Levothyroxin
Drug: Placebo
  Arms: Placebo

SUMMARY:
Hypothyroidism is risk factor in atherosclerotic cardiovascular diseases, but there is a controversy in effect of subclinical hypothyroidism on cardiovascular diseases. We aim to estimate the relation between subclinical hypothyroidism and endothelial dysfunction and the effects of levothyroxine therapy on it. Patients with confirmed subclinical hypothyroidism by lab results will be randomized to two groups of treatment with one daily dose of 100 mg Levothyroxine or placebo. The flow-mediated dilation and intima media thickness are evaluated before and after the study.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 65
* confirmed subclinical hypothyroidism

Exclusion Criteria:

* receiving of other treatments for hypothyroidism
* patients with other major medical disorders
* smoking
* hyperlipidemia
* obesity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-05; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline flow-mediated dilation at 2 months | At baseline and then 2 months after treatment
  Flow-mediated dilation will be assessed using standard method with a radiologist unaware to the study arms at baseline and then 2 months after treatment.
Change from baseline intima-media thickness at 2 months | At baseline and then 2 months after treatment
  Intima-media thickness will be assessed using standard method with a radiologist unaware to the study arms at baseline and then 2 months after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Nasmi Niknam, M.D., Principal Investigator — Isfahan University of Medical Sciences
Locations (1):
- Khorshid endocrinology clinic, Isfahan, Isfahan, Iran

REFERENCES:
- [Background] Walsh JP, Bremner AP, Bulsara MK, O'Leary P, Leedman PJ, Feddema P, Michelangeli V. Subclinical thyroid dysfunction as a risk factor for cardiovascular disease. Arch Intern Med. 2005 Nov 28;165(21):2467-72. doi: 10.1001/archinte.165.21.2467. PMID 16314542
- [Background] Alibaz Oner F, Yurdakul S, Oner E, Kubat Uzum A, Erguney M. Evaluation of the effect of L-thyroxin therapy on endothelial functions in patients with subclinical hypothyroidism. Endocrine. 2011 Oct;40(2):280-4. doi: 10.1007/s12020-011-9465-2. Epub 2011 Apr 20. PMID 21505892